CLINICAL TRIAL: NCT01641913
Title: Determination of Intestinal Permeability and Response to Treatment in Patients With Eosinophilic Esophagitis
Brief Title: Intestinal Permeability in Response to Treatment in Eosinophilic Esophagitis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Katzka, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-001344
Record Dates: First submitted 2012-07-10; First posted 2012-07-17 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Absorbable sugars (Experimental): Lactulose (1,000 mg) and mannitol (200 mg). For the liquid formulation, these sugars will be administered in 250 ml of water. After oral ingestion of the sugars in liquid form, urine will be collected every 30 minutes for the first 2 hours.
  Interventions: Other: Absorbable sugars

INTERVENTIONS:
Other: Absorbable sugars — Lactulose (1,000 mg) and mannitol (200 mg). For the liquid formulation, these sugars will be administered in 250 ml of water. After oral ingestion of the sugars in liquid form, urine will be collected every 30 minutes for the first 2 hours.

SUMMARY:
Do patient's with eosinophilic esophagitis have increased small intestinal permeability and if this changes in response to topically administered esophageal steroids?

DETAILED DESCRIPTION:
Eosinophilic esophagitis is an allergy mediated disease in which antigens exposed to the gastrointestinal tract trigger a combined immediate hypersensitivity.

The investigators anticipate that patients with active eosinophilic esophagitis will have increased intestinal permeability on urine collection of sugars. The investigators are not sure whether these findings will be found in patients who have been successfully treated with topical esophageal steroids. Improvement in intestinal permeability would be perceived as indicating that esophageal disease drives the intestinal permeability. Lack of improvement would indicate that eosinophilic esophagitis is a more systemic disease in which increased small bowel permeability is a marker or perhaps important driver of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 18 and 80 with Eosinophilic Esophagitis diagnosed by compatible symptoms, endoscopic findings, histology and lack of response to proton pump inhibitors or negative pH study.

Exclusion:

* Vulnerable populations, such as those with diminished mental acuity, will be excluded.
* Patients allergic to Lactulose
* Women who are pregnant or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To assess patients gastrointestinal symptoms in patients with EoE by means of standard validated questionnaires | 30 days
  heartburn, trouble swallowing

SECONDARY OUTCOMES:
To determine if patients with eosinophilic esophagitis have increased small intestinal permeability and if this changes in response to topically administered esophageal steroids. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: David Katzka, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States